CLINICAL TRIAL: NCT00036881
Title: Phase III Double-Blind, Placebo-Controlled Randomized Comparison Of Zinc Sulfate Versus Placebo For The Prevention Of Altered Taste In Patients With Head And Neck Cancer During Radiation
Brief Title: Zinc Sulfate in Preventing Loss of Sense of Taste in Patients Undergoing Radiation Therapy for Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N01C4; NCI-2012-02465 (Registry Identifier: CTRP (Clinical Trials Reporting System)); NCI-P02-0224; CDR0000069337 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-05-13; First posted 2003-01-27 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Dysgeusia; Head and Neck Cancer; Oral Complications; Radiation Toxicity
MeSH Terms: conditions — Dysgeusia; Head and Neck Neoplasms; Radiation Injuries | interventions — Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- zinc sulfate (Experimental): Patients receive oral zinc sulfate 3 times daily beginning the first week of radiotherapy.
  Treatment continues daily during and for 1 month after radiotherapy in the absence of unacceptable toxicity.
  Quality of life is assessed at baseline, weekly during treatment, and then at 1, 2, 3, and 6 months after the completion of treatment.
  Patients are followed at 1, 2, 3, and 6 months after the completion of treatment and then every 6 months for 1 year.
  Interventions: Dietary Supplement: zinc sulfate
- placebo (Placebo Comparator): Patients receive oral placebo 3 times daily beginning the first week of radiotherapy.
  Treatment continues daily during and for 1 month after radiotherapy in the absence of unacceptable toxicity.
  Quality of life is assessed at baseline, weekly during treatment, and then at 1, 2, 3, and 6 months after the completion of treatment.
  Patients are followed at 1, 2, 3, and 6 months after the completion of treatment and then every 6 months for 1 year.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: zinc sulfate
  Arms: zinc sulfate
Other: placebo
  Arms: placebo

SUMMARY:
RATIONALE: It is not yet known whether zinc sulfate is effective in preventing the loss of ability to taste food in cancer patients who are undergoing radiation therapy for head and neck cancer.

PURPOSE: Randomized phase III trial to determine the effectiveness of zinc sulfate in preventing loss of sense of taste in patients who are undergoing radiation therapy for head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether zinc sulfate prolongs the time to onset of altered taste in patients with head and neck cancer undergoing radiotherapy.
* Determine whether this drug decreases the overall incidence of altered taste in these patients.
* Determine whether this drug results in fewer radiotherapy treatment interruptions in these patients.
* Assess the quality of life of patients treated with this drug.
* Determine the toxic effects of this drug in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to planned radiotherapy dose (less than 6,000 cGy vs at least 6,000 cGy), estimated amount of oral mucosa in the radiation field (60% or less vs more than 60%), age (under 50 vs 50 and over), concurrent chemotherapy (yes vs no), and smoking (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral zinc sulfate 3 times daily beginning the first week of radiotherapy.
* Arm II: Patients receive oral placebo 3 times daily beginning the first week of radiotherapy.

Treatment in both arms continues daily during and for 1 month after radiotherapy in the absence of unacceptable toxicity.

Quality of life is assessed at baseline, weekly during treatment, and then at 1, 2, 3, and 6 months after the completion of treatment.

Patients are followed at 1, 2, 3, and 6 months after the completion of treatment and then every 6 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of head and neck cancer
* No stage I laryngeal cancer
* Planned treatment with at least 2,000 cGy of external beam radiotherapy to at least 30% of the oral cavity

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Gastrointestinal:

* Able to tolerate oral medication
* No known mechanical obstruction of the alimentary tract
* No malabsorption
* No intractable vomiting (more than 5 episodes per week)

Other:

* No known intolerance to zinc sulfate
* No known, untreated oral thrush
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Surgery:

* No prior surgery that included ablation or removal of the olfactory component of taste

Other:

* No concurrent zinc supplements

  * Concurrent standard multivitamins allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2002-05; Primary Completion 2007-04 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Prolongation of the time to onset of altered taste by zinc sulfate | Up to 1.5 years

SECONDARY OUTCOMES:
Incidence of taste alteration | Up to 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Study Chair — Mayo Clinic

REFERENCES:
- [Result] Halyard MY, Jatoi A, Sloan JA, Bearden JD 3rd, Vora SA, Atherton PJ, Perez EA, Soori G, Zalduendo AC, Zhu A, Stella PJ, Loprinzi CL. Does zinc sulfate prevent therapy-induced taste alterations in head and neck cancer patients? Results of phase III double-blind, placebo-controlled trial from the North Central Cancer Treatment Group (N01C4). Int J Radiat Oncol Biol Phys. 2007 Apr 1;67(5):1318-22. doi: 10.1016/j.ijrobp.2006.10.046. PMID 17394940